CLINICAL TRIAL: NCT05795400
Title: Administration of the SGLT-2 Inhibitor Dapagliflozin in the Patients With Amyloid Cardiomyopathy: a Pilot Study
Brief Title: Administration of the SGLT-2 Inhibitor Dapagliflozin in the Patients With Amyloid Cardiomyopathy
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Medical Research Center for Cardiology, Ministry of Health of Russian Federation (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20230120
Record Dates: First submitted 2023-01-20; First posted 2023-04-03 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-02

CONDITIONS: Heart Failure With Reduced Ejection Fraction; Heart Failure With Preserved Ejection Fraction; Heart Failure With Mid Range Ejection Fraction; Amyloid Cardiomyopathy
Keywords: heart failure; amyloidosis; cardiomyopathy; amyloid cardiomyopathy
MeSH Terms: conditions — Amyloid Neuropathies, Familial; Heart Failure; Amyloidosis; Cardiomyopathies | interventions — dapagliflozin

STUDY DESIGN:
Intervention Model Description: a single-center, pilot, prospective, randomized, placebo-controlled clinical trial
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dapagliflozine group (Experimental): 20 patients diagnosed with heart failure and amyloid cardiomyopathy, regardless of HF phenotype, are planned to be enrolled in the study. Patients with the edematous syndrome are allowed to participate in the study, but the condition of stable hemodynamics must be observed. Regardless of the group, patients will receive standard therapy for ADHF (diuretics and MRA). Patients will not receive beta-blockers/ACE-I/ARNI. In the treatment group the therapy will include the SGLT-2 inhibitor dapagliflozin, which will be prescribed during the first 24 hours after the hospitalization.
  Interventions: Drug: Dapagliflozin 10mg Tab
- Control group (Placebo Comparator): In the control group, patients will be treated with standard diuretic therapy without SGLT-2 inhibitors.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dapagliflozin 10mg Tab — 10 mg tablets given once daily, per oral use
  Arms: Dapagliflozine group
Drug: Placebo — tablet of placebo drug dosed once daily
  Arms: Control group

SUMMARY:
Efficacy and safety of early administration of the SGLT-2 inhibitor dapagliflozin will be evaluated in patients with HF, regardless of LVEF, due to amyloid cardiomyopathy.

DETAILED DESCRIPTION:
Amyloidosis is an infiltrative disease in which fibrillar glycoprotein amyloid is deposited in the tissues. The prevalence of amyloidosis remains largely unexplored, but if the wild type of transthyretin amyloidosis is considered, it still remains significantly underestimated in the population. Among patients hospitalized for heart failure with a preserved left ventricular ejection fraction (HFpEF), 13% are later diagnosed with amyloid cardiomyopathy (AC), in 20-25% of patients over 80 years old AC is a finding of pathologists, and in the oldest group of patients over 97 years old AC is identified in 37% of cases. Hereditary transthyretin amyloidosis occurs at less than 8.8 cases per 1 million population in non-endemic areas (e.g., Sicily) and 1 case per 1000 population in endemic areas (e.g., Portugal). Thus, the prevalence of amyloid cardiomyopathy as the cause of HFpEF is underestimated.

One of the manifestations of systemic amyloidosis is amyloid cardiomyopathy, when amyloid is deposited in the myocardium. This leads to thickening walls (phenotype of hypertrophic cardiomyopathy) and impaired relaxation processes, leading to diastolic myocardial dysfunction up to restrictive disorders (restrictive cardiomyopathy phenotype). Thus, in patients with amyloid cardiomyopathy HFpEF develops, and with the progression of the disease - heart failure with the mildly reduced (HFmrEF) and reduced (HFrEF) ejection fraction. The tragedy of situation lies in the fact that the specific (disease-modifying) treatment aimed at stopping or delaying amyloid deposition is limited to only two types of amyloidosis: AL and ATTR. As for the symptomatic treatment of HF, unfortunately, according to specific changes in hemodynamics, even with the reduced LVEF, therapy with beta-blockers, ACE-I/ARB/ARNI should be canceled. Currently, with the manifestation of the symptoms of HF, strict control over the drinking regimen and hydrobalance is necessary, and salt intake should be limited. In case of oedema, treatment with loop diuretics, MRA should be administrated. To date, in the treatment of HF, both with the reduced and preserved LVEF, another group of drugs has appeared - sodium-glucose cotransporter-2 (SGLT-2) inhibitors. However, in all studies conducted, the presence of HCM/RCM was the non-inclusion criteria in the investigation. At the same time, this group of drugs, unlike beta-blockers/ACE-I/ARNI, doesn't have such a significant effect on central hemodynamics, but it can have a positive antiproliferative, metabolic and nephroprotective effect.

Thereby, the study of SGLT-2 use in patients with amyloid cardiomyopathy with any phenotype of HF compared to placebo is of special interest.

Aims: Determination of the possibility of influence of early administration of SGLT-2 inhibitor dapagliflozin on a course of the disease (functional status, clinical and laboratory parameters, systolic and diastolic function of the left and right ventricular, cardiac strain parameters, parameters of target organ functions) in patients with the acute decompensated heart failure (ADHF), regardless of LVEF, against the background of transthyretin amyloid cardiomyopathy.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females between 18 and 80 years of age
2. HF, confirmed with the increased level of NT-proBNP>300 pg/mL or BNP>100 pg/mL
3. Transthyretin amyloid cardiomyopathy, confirmed with echocardiography and/or contrast-enhanced cardiac MRI

Exclusion Criteria:

1. The inability to continue all the activities planned in this study by the patient.
2. The onset of pregnancy.
3. Patient's voluntary withdrawal of consent to participate in a clinical trial at any point during the conduct of the study.
4. Development of intolerable side effects.
5. Administration of disease-modifying treatment of amyloidosis.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2025-02-26 (Actual); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Effect of dapagliflozin on quality of life using Kansas City Cardiomyopathy Questionnaire Summary Score (KCCQ-SC) | 6 months
  Changes in KCCQ score will be assessed
Effect of Dapagliflozin on 6 Minute Walk Test Distance | 6 months
  Changes in 6MWT score will be assessed
Effect of dapagliflozin on N-terminal Pro B-type Natriuretic Peptide (NTproBNP) | 6 months
  Changes in concentration of NT-proBNP will be assessed

SECONDARY OUTCOMES:
Cardiovascular death + number of hospitalizations due to heart failure | 6 months
Effect of dapagliflozin on change in echocardiographic parameters | 6 months
  Left ventricular ejection fraction will be assessed
Effect of dapagliflozin on change in specle-tracking echocardiographic parameters | 6 months
  Global longitudinal strain will be assessed

CONTACTS AND LOCATIONS:
Locations (1):
- National Medical Research Center for Cardiology, Ministry of Health of Russian Federation, Moscow, Russia

IPD SHARING:
Plan to Share IPD: Undecided